CLINICAL TRIAL: NCT02657031
Title: The Check Trial: A Comparison of Headache Treatment in the ED: Compazine Versus Ketamine. A Multi-Center, Randomized Double-Blind, Clinical Control Trial.
Brief Title: The CHECK Trial: A Comparison of Headache Treatment in the ED: Compazine Versus Ketamine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Medical Center of Southern Nevada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EM 2015.13
Record Dates: First submitted 2016-01-13; First posted 2016-01-15 (Estimated); Results first posted 2017-12-11 (Actual); Last update posted 2017-12-11 (Actual); Status verified 2017-12

CONDITIONS: Headache
Keywords: Headache, Migraine
MeSH Terms: conditions — Headache; Migraine Disorders | interventions — Prochlorperazine; Ketamine; Diphenhydramine; Ondansetron; Saline Solution

STUDY DESIGN:
Intervention Model Description: Double-Blind Randomized Clinical Control Trial
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Arm (Active Comparator): This arm uses standard of care treatment of prochlorperazine 10 mg IV along with diphenhydramine 25 mg IV plus Normal Sailine 500 cc bolus
  Interventions: Drug: Prochlorperazine; Drug: Diphenhydramine; Drug: Normal Saline
- Study Arm (Experimental): This arm uses stud drug regime of Ketamine 0.3 mg/kg along with Ondansetron 4 mg IV plus Normal Saline 500 cc bolus.
  Interventions: Drug: Ketamine; Drug: Ondansetron; Drug: Normal Saline

INTERVENTIONS:
Drug: Prochlorperazine — prochlorperazine 10 mg IV
  Other Names: Compazine
  Arms: Control Arm
Drug: Ketamine — Ketamine 0.3 mg/kg IV
  Other Names: Ketalar
  Arms: Study Arm
Drug: Diphenhydramine — Diphenhydromine 25 mg IV
  Other Names: Benadryl
  Arms: Control Arm
Drug: Ondansetron — Ondansetron 4 mg IV
  Other Names: Zofran
  Arms: Study Arm
Drug: Normal Saline — Normal Saline 500 cc IV Bolus
  Other Names: NS

SUMMARY:
This study compares the efficacy of low dose Ketamine versus Compazine for the control of headache in patients presenting to the Emergency Department.

DETAILED DESCRIPTION:
After enrollment, each patient will randomized either to the standard treatment arm to receive prochlorperazine 10 mg IV along with diphenhydramine 25 mg IV, OR to the study arm to receive Ketamine 0.3 mg/kg along with ondansetron 4 mg IV. The diphenhydramine or ondansetron will be administered first, and immediately afterward the prochlorperazine or Ketamine will be administered. The prochlorperazine or Ketamine will be diluted in saline so that the total volume is 5 mL, and will be administered over 2 minutes. The diphenhydramine will be diluted in saline so that it is 2 mL (the same volume as the ondansetron). Both groups will also receive a 500 mL normal saline bolus after the study medications are administered. The ED pharmacist will be responsible for preparing the medications, using a double-blind protocol. He or she will record which arm the patient was randomized to. Only the pharmacist will have access to the randomization records and will not reveal the randomization until the end of the study. Emergency providers will be instructed not to administer any rescue medications for at least 30 minutes. The electronic medical record order will read "randomized study medication" (for the Ketamine or prochlorperazine) and "randomized add-on medication" (for the ondansetron or diphenhydramine).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years
* Temperature < 100.4° F
* Diastolic Blood Pressure <104 mm Hg
* Normal neurological exam and mormal mental status

Exclusion Criteria:

* Pregnant or breastfeeding.
* Meningeal signs are present
* Acute angle closure glaucoma is suspected.
* Head trauma within the previous two weeks
* Lumbar puncture within the previous two weeks
* Thunderclap onset of the headache
* Weight more than 150 kg or less than 40 kg.
* Known allergy to one of the study drugs.
* History of schizophrenia or bipolar disorder.
* History of intracranial hypertension.
* Is a prisoner
* Patient declined informed consent
* Non-English speaking patient.
* Attending provider excludes patient

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-03-17 (Actual); Primary Completion 2017-03-21 (Actual); Study Completion 2017-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A Zitek, MD, Principal Investigator — Unviersity of Nevada School of Medicine
Locations (1):
- University Medical Center of Southern Nevada, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No
This was intended a multi-center (2 sites) study that would have shared redacted data with investigators from both sites, however, site #2 did not receive a data sharing agreement or IRB approval from their institution. So by default the study effectively became a single site study.

REFERENCES:
- [Result] Pitts SR, Niska RW, Xu J, Burt CW. National Hospital Ambulatory Medical Care Survey: 2006 emergency department summary. Natl Health Stat Report. 2008 Aug 6;(7):1-38. PMID 18958996
- [Result] Gelfand AA, Goadsby PJ. A Neurologist's Guide to Acute Migraine Therapy in the Emergency Room. Neurohospitalist. 2012 Apr 1;2(2):51-59. doi: 10.1177/1941874412439583. PMID 23936605
- [Result] Cicek M, Karcioglu O, Parlak I, Ozturk V, Duman O, Serinken M, Guryay M. Prospective, randomised, double blind, controlled comparison of metoclopramide and pethidine in the emergency treatment of acute primary vascular and tension type headache episodes. Emerg Med J. 2004 May;21(3):323-6. doi: 10.1136/emj.2002.000356. PMID 15107371
- [Result] Friedman BW, Adewunmi V, Campbell C, Solorzano C, Esses D, Bijur PE, Gallagher EJ. A randomized trial of intravenous ketorolac versus intravenous metoclopramide plus diphenhydramine for tension-type and all nonmigraine, noncluster recurrent headaches. Ann Emerg Med. 2013 Oct;62(4):311-318.e4. doi: 10.1016/j.annemergmed.2013.03.017. Epub 2013 Apr 6. PMID 23567060
- [Result] Kostic MA, Gutierrez FJ, Rieg TS, Moore TS, Gendron RT. A prospective, randomized trial of intravenous prochlorperazine versus subcutaneous sumatriptan in acute migraine therapy in the emergency department. Ann Emerg Med. 2010 Jul;56(1):1-6. doi: 10.1016/j.annemergmed.2009.11.020. Epub 2010 Jan 4. PMID 20045576
- [Result] Tanen DA, Miller S, French T, Riffenburgh RH. Intravenous sodium valproate versus prochlorperazine for the emergency department treatment of acute migraine headaches: a prospective, randomized, double-blind trial. Ann Emerg Med. 2003 Jun;41(6):847-53. doi: 10.1067/mem.2003.195. PMID 12764341
- [Result] Jones J, Sklar D, Dougherty J, White W. Randomized double-blind trial of intravenous prochlorperazine for the treatment of acute headache. JAMA. 1989 Feb 24;261(8):1174-6. PMID 2915441
- [Result] Friedman BW, Esses D, Solorzano C, Dua N, Greenwald P, Radulescu R, Chang E, Hochberg M, Campbell C, Aghera A, Valentin T, Paternoster J, Bijur P, Lipton RB, Gallagher EJ. A randomized controlled trial of prochlorperazine versus metoclopramide for treatment of acute migraine. Ann Emerg Med. 2008 Oct;52(4):399-406. doi: 10.1016/j.annemergmed.2007.09.027. Epub 2007 Nov 19. PMID 18006188
- [Result] Callan JE, Kostic MA, Bachrach EA, Rieg TS. Prochlorperazine vs. promethazine for headache treatment in the emergency department: a randomized controlled trial. J Emerg Med. 2008 Oct;35(3):247-53. doi: 10.1016/j.jemermed.2007.09.047. Epub 2008 Jun 5. PMID 18534808
- [Result] Coppola M, Yealy DM, Leibold RA. Randomized, placebo-controlled evaluation of prochlorperazine versus metoclopramide for emergency department treatment of migraine headache. Ann Emerg Med. 1995 Nov;26(5):541-6. doi: 10.1016/s0196-0644(95)70001-3. PMID 7486359
- [Result] Miner JR, Fish SJ, Smith SW, Biros MH. Droperidol vs. prochlorperazine for benign headaches in the emergency department. Acad Emerg Med. 2001 Sep;8(9):873-9. doi: 10.1111/j.1553-2712.2001.tb01147.x. PMID 11535479
- [Result] Friedman BW, Hochberg ML, Esses D, Grosberg BM, Rothberg D, Bernstein B, Bijur PE, Lipton RB, Gallagher EJ. Recurrence of primary headache disorders after emergency department discharge: frequency and predictors of poor pain and functional outcomes. Ann Emerg Med. 2008 Dec;52(6):696-704. doi: 10.1016/j.annemergmed.2008.01.334. Epub 2008 Apr 3. PMID 18387702
- [Result] McCarthy LH, Cowan RP. Comparison of parenteral treatments of acute primary headache in a large academic emergency department cohort. Cephalalgia. 2015 Aug;35(9):807-15. doi: 10.1177/0333102414557703. Epub 2014 Nov 3. PMID 25366551
- [Result] Adams HA. [Mechanisms of action of ketamine]. Anaesthesiol Reanim. 1998;23(3):60-3. German. PMID 9707750
- [Result] Eghbal MH, Taregh S, Amin A, Sahmeddini MA. Ketamine improves postoperative pain and emergence agitation following adenotonsillectomy in children. A randomized clinical trial. Middle East J Anaesthesiol. 2013 Jun;22(2):155-60. PMID 24180163
- [Result] Weinbroum AA. A single small dose of postoperative ketamine provides rapid and sustained improvement in morphine analgesia in the presence of morphine-resistant pain. Anesth Analg. 2003 Mar;96(3):789-795. doi: 10.1213/01.ANE.0000048088.17761.B4. PMID 12598264
- [Result] McGuinness SK, Wasiak J, Cleland H, Symons J, Hogan L, Hucker T, Mahar PD. A systematic review of ketamine as an analgesic agent in adult burn injuries. Pain Med. 2011 Oct;12(10):1551-8. doi: 10.1111/j.1526-4637.2011.01220.x. Epub 2011 Aug 31. PMID 21880111
- [Result] Hocking G, Cousins MJ. Ketamine in chronic pain management: an evidence-based review. Anesth Analg. 2003 Dec;97(6):1730-1739. doi: 10.1213/01.ANE.0000086618.28845.9B. PMID 14633551
- [Result] Andolfatto G, Willman E, Joo D, Miller P, Wong WB, Koehn M, Dobson R, Angus E, Moadebi S. Intranasal ketamine for analgesia in the emergency department: a prospective observational series. Acad Emerg Med. 2013 Oct;20(10):1050-4. doi: 10.1111/acem.12229. PMID 24127709
- [Result] Motov S, Rockoff B, Cohen V, Pushkar I, Likourezos A, McKay C, Soleyman-Zomalan E, Homel P, Terentiev V, Fromm C. Intravenous Subdissociative-Dose Ketamine Versus Morphine for Analgesia in the Emergency Department: A Randomized Controlled Trial. Ann Emerg Med. 2015 Sep;66(3):222-229.e1. doi: 10.1016/j.annemergmed.2015.03.004. Epub 2015 Mar 26. PMID 25817884
- [Result] Miner JR, Smith SW, Moore J, Biros M. Sumatriptan for the treatment of undifferentiated primary headaches in the ED. Am J Emerg Med. 2007 Jan;25(1):60-4. doi: 10.1016/j.ajem.2006.06.004. PMID 17157685

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Arm: Prochlorperazine and Diphenhydramine
- Study Arm: Ketamine and Ondansetron
Period: Overall Study
Arm/Group | Control Arm | Study Arm
Started | 29 | 25
Completed | 28 | 23
Not Completed | 1 | 2
Not completed — Adverse Event | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Control Arm: This arm uses standard of care treatment of prochlorperazine 10 mg IV along with diphenhydramine 25 mg IV plus Normal Sailine 500 cc bolus
  Prochlorperazine: prochlorperazine 10 mg IV
  Diphenhydromine: Diphenhydromine 25 mg IV
  Normal Saline: Normal Saline 500 cc IV Bolus
- Study Arm: This arm uses stud drug regime of Ketamine 0.3 mg/kg along with Ondansetron 4 mg IV plus Normal Sailing 500 cc bolus.
  Ketamine: Ketamine 0.3 mg/kg IV
  Ondansetron: Ondansetron 4 mg IV
  Normal Saline: Normal Saline 500 cc IV Bolus
- Total: Total of all reporting groups
Arm/Group | Control Arm | Study Arm | Total
Number analyzed (Participants) | 28 | 23 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 23 | 51
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.4 (10.4) | 32.3 (10.3) | 34.9 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 19 | 39
  Male | 8 | 4 | 12
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 9 | 7 | 16
Region of Enrollment [Number; unit: participants]
  United States | 28 | 23 | 51
Visual Analog Scale (VAS) Pain Score, mm [Mean (Standard Deviation); unit: mm] — Scores range from 0 mm (no pain) to 100 mm (maximum pain)
  mm | 78.3 (17.7) | 77.8 (14.6) | 78 (17)

OUTCOME MEASURES:

1. Primary Outcome: Headache Following Intervention
Description: Reduction in 100 mm Visual Analog Scale (VAS) Score. Positive values represent a reduction in headache severity. The maximum possible change in VAS score is 100 mm, representing the complete relief of a maximally severe headache. A change of 0 mm corresponds to no change in headache severity, and a negative value indicates worsening of the headache after the medication.
Time Frame: 0-60 minutes
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | Control Arm | Study Arm
Number analyzed (Participants) | 28 | 23
mm | 63.5 [52.7 to 74.3] | 43.5 [30.2 to 56.8]

2. Secondary Outcome: Anxiety
Description: Reduction in 100 mm Visual Analog Scale (VAS) Score. The maximum possible change in VAS score is 100 mm, representing the complete relief of maximum anxiety. A change of 0 mm corresponds to no change in anxiety level, and a negative value indicates worsening of the anxiety after the medication.
Time Frame: 0-60 minutes
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Control Arm | Study Arm
Number analyzed (Participants) | 28 | 23
mm | 33.7 (32.5) | 21.2 (40.5)

3. Secondary Outcome: Nausea
Description: Reduction in 100 mm Visual Analog Scale (VAS) Score. The maximum possible change in VAS score is 100 mm, representing the complete relief of maximum nausea. A change of 0 mm corresponds to no change in nausea level, and a negative value indicates worsening of the nausea after the medication.
Time Frame: 0-60 minutes
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Control Arm | Study Arm
Number analyzed (Participants) | 28 | 23
mm | 38.9 (34.8) | 22.9 (37.5)

4. Secondary Outcome: The Number of Participants Experiencing Vomiting
Description: Yes/No
Time Frame: 0-60 minutes
Measure: Number; unit: participants
Arm/Group | Control Arm | Study Arm
Number analyzed (Participants) | 28 | 23
participants | 2 | 3

5. Secondary Outcome: The Number of Patients Experiencing Restlessness
Description: Yes/No
Time Frame: 0-60 minutes
Measure: Number; unit: participants
Arm/Group | Control Arm | Study Arm
Number analyzed (Participants) | 28 | 23
participants | 3 | 3

ADVERSE EVENTS:
Time Frame: 15 minutes
Arm/Group | Control Arm | Study Arm
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/25
Other Adverse Events (participants affected / at risk) | 1/29 | 2/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Arm (N=29) | Study Arm (N=25)
Dysphoria (Nervous system disorders) | 1 (1) | 2 (2) — The patients who dropped out of the ketamine group had dysphoria; the patient who dropped out of the prochlorperazine group had akathisia

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-20): https://cdn.clinicaltrials.gov/large-docs/31/NCT02657031/Prot_SAP_000.pdf